CLINICAL TRIAL: NCT02776540
Title: Clopidogrel Loading for Acute Ischaemia of Recent Onset (CAIRO)
Brief Title: Clopidogrel for Acute Ischaemia of Recent Onset
Acronym: CAIRO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Eman Mones Abushady, Assistant Lecturer of Neurology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAIRORCT
Record Dates: First submitted 2016-05-02; First posted 2016-05-18 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Ischemic Cerebrovascular Accident
MeSH Terms: conditions — Ischemic Stroke | interventions — Clopidogrel; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 900 mg Clopidogrel (Active Comparator): 67 patients will receive 12 tablets clopidogrel ( each 75 mg) as total 900 mg each patient
  Interventions: Drug: Clopidogrel
- 600 mg Clopidogrel (Active Comparator): 67 patient will receive 8 tablets clopidogrel (each 75 mg) as total 600 mg each patient and 4 tablets placebo to receive 12 tablets as total
  Interventions: Drug: Clopidogrel
- 400 mg Aspirin (Placebo Comparator): 67 patients will receive 4 tablets Aspirin ( each 75 mg) as total 300 mg for each patient and 8 tablets placebo to receive 12 tablets as total
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Clopidogrel — there is 2 groups one group will receive 900 mg Clopidogrel and the other will receive 600 mg Clopidogrel
  Other Names: Srtoka
  Arms: 600 mg Clopidogrel; 900 mg Clopidogrel
Drug: Aspirin — there's another group will receive 400 mg Aspirin
  Other Names: Aspocid
  Arms: 400 mg Aspirin

SUMMARY:
Evaluate the role of loading Clopidogrel in acute ischemic stroke in improving neurological outcome of stroke in cases patients will be non-eligible for, or declined, treatment with or intravenous thrombolysis with rTPA, rTPA is not available or thrombectomy.

ELIGIBILITY:
Inclusion Criteria:

1. First ever presentation with acute ischemic stroke. Previous transient ischemic attacks (TIA's) are not excluding, regardless of their frequency or severity
2. Ictus to drug time does not to exceed 9 hours (allowing for at least 30 minutes to obtain imaging)
3. Patients with undetermined time of onset will be included only if they were last seen well within the same time window (9hrs). Onset of events in patients presented with stuttering stroke will be considered from the onset of the first clinical manifestation.
4. According to National Institute of Health Stroke Scale (NIHSS) on admission, patient will be recruited with NIHSS between 4 and 24 (both inclusive).

Exclusion Criteria:

1. Patients eligible for intravenous (recombinant tissue plasminogen activator) rTPA thrombolysis or thrombectomy.
2. If NIHSS on admission is 3 or less, 25 or more, or patients who are showing rapidly resolving symptoms prior to the results of imaging.
3. Clinical seizures at the onset of stroke.
4. Patients with known history or manifestations of any major organ failure.
5. Patients who have had acute myocardial infarction within 1 month; and/or with management interfering with the current study (e.g. warfarin).
6. Patients with active malignancies, and/or have been on chemo- or radiotherapy within the last year.
7. Patients with active peptic ulcer and/or (gastrointestinal tract) GIT surgery or bleeding within the last year.
8. Persistent uncontrolled vomiting during the first day of admission.
9. Patients with major surgery within the last 3 months.
10. Patients with history of uncontrolled bleeding site, within the prior year.
11. Patients with known allergy to study drugs.
12. Patients with known history of persistent or recurrent (central nervous system) CNS pathology (e.g. epilepsies, meningioma, multiple sclerosis).
13. Patients with past history of head trauma with residual neurological deficit
14. Patients who are on regular Clopidogrel during the week before admission.
15. Patient with raised prothrombin time (PT) on admission, either on anticoagulants (with raised INR>1.3, PT >18 second) or not (PT> 15 second), or on drugs that might increase possibility of peripheral bleeding (e.g. corticosteroids).
16. Patients who have an indication for full anti-coagulation during the first week of their hospital stay will be retrospectively excluded.
17. Patients receiving anti-coagulants in deep venous thrombosis (DVT) prophylaxis doses will NOT be excluded:

    * Enoxaparin 40mg/d (or equivalent).
    * Heparin with partial thromboplastin time (PTT) not exceeding 50 seconds.
    * Oral anticoagulation with INR <1.5.
18. Pregnancy or breast feeding
19. Stroke due to venous thrombosis
20. Hemorrhagic stroke
21. Blood pressure < 90/60 or > 185/110 mmHg, if not responding to intravenous antihypertensive therapy or requiring aggressive treatment to reduce it below this limit
22. Arterial puncture in a non-compressible site within the previous week
23. Strokes following cardiac arrest or profuse hypotension.
24. Blood glucose level < 50 or > 400 mg/dl on admission
25. CBC with picture of severe anemia (Haematocrit <0.25), thrombocytopenia (Platelets < 100,000) or leucopenia (WBC < 3,000).
26. Significant electrolyte imbalance that may account for the presenting manifestations
27. Contraindications to imaging
28. Urgent brain CT revealing any of the following:

    * Hemorrhage.
    * Major cerebral non-vascular pathology.
    * Suspected arterio-venous malformation (AVM).
    * Previous intracerebral hemorrhage or old infarctions larger than 1.5 cm.
    * Massive acute hypo density in the brain region corresponding to the current symptoms.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
The change of NIH stroke scale score | Baseline and up to 1 week
  Patients will be assessed for early neurologic improvement or deterioration using the change of NIH stroke scale score. Early neurological outcome
Neurologic outcome | 3 months
  patients will be assessed for neurologic outcome using the Modified Ranking Scale at 3 months after onset

SECONDARY OUTCOMES:
Bleeding complications of loading clopidogrel | 1 week
  will follow cerebral bleeding complications using CT scan, and systemic bleeding complications (GI bleeding, hematuria, etc.) that may occur following the loading dose

CONTACTS AND LOCATIONS:
Overall Officials: Ramez R Moustafa, MD PhD MRCP, Principal Investigator — Department of Neurology, Ain Shams University
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt